CLINICAL TRIAL: NCT06248684
Title: Prevention of Postoperative Delirium in the Care of Elderly Patients. A Monocentric, Prospective Intervention Study
Brief Title: Prevention of Postoperative Delirium in Elderly Patients
Acronym: PODproject
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Postoperative delirium project
Record Dates: First submitted 2023-10-01; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Delirium
Keywords: delirium, prevention and control; post operative delirium; delirium, risk factors; delirium, risk assessment; Baseline-EEG; cognitive tests; EEG, intraoperative
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prevention group (Other): patients receive standardized perioperative care using Standard Operating Procedures (SOPs) in accordance with the guidelines of the professional societies for the prevention of postoperative delirium.
  Interventions: Other: standardized prevention and therapy measures

INTERVENTIONS:
Other: standardized prevention and therapy measures — Patients from the age of 65 years with an additional risk factor for postoperative delirium are assigned to a multidimensional standardized perioperative care protocol.

SUMMARY:
Prevention of Postoperative Delirium in the care of Elderly Patients. A Monocentric, Prospective Intervention Study With the Question of Whether the Incidence, Length and Severity of Postoperative Delirium Can be Reduced by Implementing a Standardised, Multidimensional Delirium Management Protocol.

DETAILED DESCRIPTION:
Within the framework of a six-month observation period, the investigators intend to identify risk factors of the patient collective for the development of postoperative delirium. For this purpose, a preoperative risk assessment is performed, which includes cognitive and physical performance as well as premedication and concomitant diseases. Included are patients of at least 65 years of age of defined specialties. Postoperatively, patients who have undergone the assessment are tested for delirium once per shift until the third postoperative day and severity and duration are documented. After completion of the observation period, risk factors favoring the development of postoperative delirium will be identified. In the subsequent intervention period, patients from the age of 65 years with an additional identified risk factor will receive standardized, targeted perioperative care. This includes both adherence to preventive measures in accordance with guidelines and the recommendation of therapeutic measures if a delirium is diagnosed. Through the standardized, interprofessional and interdisciplinary application of the described approach, the investigator aim to reduce the incidence, duration and severity of postoperative delirium. Furthermore, the evaluation of the identification of the weighting of risk factors as well as the identification of risk factors by the tests performed, length of hospital stay, three-month mortality and daily living skills after three months. In addition, a baseline EEG (standardized awake EEG before initiation) is recorded in a subgroup to determine whether patients at risk for delirium can be identified and whether intraoperative EEG parameters support the delirium risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 Years
* intervention in one of the following departments: general and visceral surgery, urology, vascular surgery, orthopedics, trauma surgery,
* Written consent by patient or legal guardian

Exclusion Criteria:

* Foreign language patients without interpreter
* non-consenting patients without a legal representative

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2024-02-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | for three days postoperatively and if the patient is delirium positive on the last day for the period until he is delirium negative or discharged from inpatient care, up to the day 90 visit at the latest
  Patients are examined once per shift for the described duration postoperatively using validated tests for delirium (CAM-ICU or 3D-CAM). Delirium testing is supplemented by pain assessment using the numerical rating scale (NRS).

SECONDARY OUTCOMES:
duration of postoperative delirium | for three days postoperatively and if the patient has delirium on the last day for the period until he is delirium negative or discharged from inpatient care, up to the day 90 visit at the latest
  Patients are examined once per shift for the described duration postoperatively using validated tests for delirium (CAM-ICU or 3D-CAM). Delirium testing is supplemented by pain assessment using the numerical rating scale (NRS).
Severity of the postoperative delirium | for three days postoperatively and if the patient has delirium on the last day for the period until he is delirium negative or discharged from inpatient care, up to the day 90 visit at the latest
  Patients are examined once per shift for the described duration postoperatively using validated tests for delirium severity (CAM-ICU or 3D-CAM). Delirium testing is supplemented by pain assessment using the numerical rating scale (NRS).
Which parameters and tests detect patients at risk for postoperative delirium? | From the time of premedication until three days postoperatively
  analysis of the preoperative risk assessment, perioperative clinical parameters and postoperative delirium screening.
Can baseline and intraoperative EEG parameters be used to identify patients at risk? Does intraoperative burst suppression EEG represent a risk factor for delirium? | From the patient's arrival in the operating room to three days postoperatively
  Analysis of EEG data recorded immediately before induction of anesthesia and during surgery.
When is the diagnosis of postoperative delirium most commonly made? | for three days postoperative
  Patients are examined once per shift for the described duration postoperatively using validated tests for delirium (CAM-ICU or 3D-CAM). Delirium testing is supplemented by pain assessment using the numerical rating scale (NRS).
The implementation of a delirium management protocol during the intervention period serves to improve the three-month outcome of patients at risk in terms of maintaining their autonomy or daily living skills. | One-time interview three months postoperatively
  Patients are asked about their daily living skills by telephone three months after their surgical procedure.
Implementation of a delirium management protocol reduces the length of hospital stay of risk patients | from the date of hospitalisation to the date of discharge from hospital, up to the day 90 visit at the latest
  The length of inpatient stay of patients before and after implementation of standardized care is evaluated
Implementation of a delirium management protocol reduces three-month mortality in high-risk patients | Query of the patients' death data three months postoperatively
  Three-month mortality of patients before and after implementation of standardized care is evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prof. Dr. med. Schneider, MD, Principal Investigator — clinic for anesthesiology and intensive care, Klinikum rechts der Isar, Technical University Munich

IPD SHARING:
Plan to Share IPD: No